CLINICAL TRIAL: NCT02710123
Title: Sub-Threshold Exercise Treatment for Adolescents With Sports Related Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, John Leddy, Principal Investigator, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 030-690120; UL1TR001412 (NIH)
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Brain Injury; Concussion
MeSH Terms: conditions — Brain Injuries; Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise (Experimental): Participants will receive an exercise prescription based on their heart rate threshold (HRT) for symptom exacerbation during the Buffalo Concussion Treadmill Test (BCTT). The script will ask the participant to exercise one a day for 20 minutes at 80% of HRT. Participants will wear a smart watch to monitor their frequency, actual time and HR during exercise. Treatment will continue until participant is fully recovered from their concussion. Intervention: Sub-Threshold exercise prescription
  Interventions: Other: Sub-Threshold exercise prescription
- Stretching Exercise (Placebo Comparator): Participants will receive a prescription for stretching exercises that they will be asked to do daily. Participants will wear a smart watch to monitor their frequency, actual time and HR during exercise. Treatment will continue until participant is fully recovered from their concussion. Intervention: Structured stretching exercise prescription.
  Interventions: Other: Structured stretching prescription

INTERVENTIONS:
Other: Sub-Threshold exercise prescription — Participants will be given a prescription to exercise at 80% of their threshold HR for symptom exacerbation. HR Threshold will be monitored weekly and exercise level increased accordingly.
  Arms: Aerobic Exercise
Other: Structured stretching prescription — Participants will be given a prescription for daily stretching lasting approximately 20 minutes.
  Arms: Stretching Exercise

SUMMARY:
Adolescents with concussion will be randomly assigned to a treatment group where they will receive sub-threshold exercise, or assigned to a placebo group where they will receive structured stretching exercises. Both groups will receive standard medical coverage with regular clinic visits. All participants will record symptoms daily on a dedicated web site. All participants will be evaluated at time 1 with (1) structured physical exam, and (2) structured exercise stress test which is terminated when there is symptom exacerbation. The primary outcome measure is time to recovery where recovery is defined as (1) asymptomatic for two consecutive days, and (2) ability to exercise to exhaustion without exacerbation of symptoms, and (3) confirmed by a physician based on a structured physical exam.

DETAILED DESCRIPTION:
Adolescents with concussion will be randomly assigned to a treatment group where they will receive sub-threshold exercise, or assigned to a placebo group where they will receive structured stretching exercises. Both groups will receive standard medical coverage with regular clinic visits. All participants will record symptoms daily on a dedicated web site. All participants will be evaluated at time 1 with (1) structured physical exam, and (2) structured exercise stress test which is terminated when there is symptom exacerbation. The primary outcome measure is time to recovery where recovery is defined as (1) asymptomatic for two consecutive days, and (2) ability to exercise to exhaustion without exacerbation of symptoms, and (3) confirmed by a physician based on a structured physical exam.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent with concussion injury from sports within first 10 days

Exclusion Criteria:

* Evidence of focal neurologic deficit; ADHD; history of moderate or severe TBI; greater than 3 prior concussions (or having history of long recovery from concussion, >3 mths); inability to understand English

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Leddy, MD, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Derived] Castellana MC, Burnett GJ, Gasper A, Nazir MSZ, Leddy JJ, Master CL, Mannix RC, Meehan WP 3rd, Willer BS, Haider MN. Adolescents With a High Burden of New-Onset Mood Symptoms After Sport-Related Concussion Benefit From Prescribed Aerobic Exercise, a Secondary Analysis of 2 Randomized Controlled Trials. Clin J Sport Med. 2025 Jan 1;35(1):29-36. doi: 10.1097/JSM.0000000000001242. Epub 2024 Jul 9. PMID 38980666
- [Derived] Willer BS, Haider MN, Bezherano I, Wilber CG, Mannix R, Kozlowski K, Leddy JJ. Comparison of Rest to Aerobic Exercise and Placebo-like Treatment of Acute Sport-Related Concussion in Male and Female Adolescents. Arch Phys Med Rehabil. 2019 Dec;100(12):2267-2275. doi: 10.1016/j.apmr.2019.07.003. Epub 2019 Aug 1. PMID 31377190
- [Derived] Leddy JJ, Haider MN, Ellis MJ, Mannix R, Darling SR, Freitas MS, Suffoletto HN, Leiter J, Cordingley DM, Willer B. Early Subthreshold Aerobic Exercise for Sport-Related Concussion: A Randomized Clinical Trial. JAMA Pediatr. 2019 Apr 1;173(4):319-325. doi: 10.1001/jamapediatrics.2018.4397. PMID 30715132

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 165 eligible candidates, 113 were randomized, 10 were lost to follow-up and 103 were included in the analysis.
Period: Overall Study
Arm/Group | Aerobic Exercise | Stretching Exercise
Started | 57 | 56
Completed | 52 | 51
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Illness unrelated to study intervention | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise | Stretching Exercise | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age
  Years | 15.3 (1.6) | 15.4 (1.7) | 15.3 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 31 | 30 | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  United States | 57 | 56 | 113
Time since injury [Median (Standard Deviation); unit: Days] | 4.9 (2.2) | 4.8 (2.4) | 4.9 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Time (in Days) to Recovery
Description: Time (in days) to recovery (Recovery is asymptomatic+able to exercise to exhaustion without symptom exacerbation+judged recovered by MD with structured physical exam.)
Time Frame: 2 to 180 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Aerobic Exercise | Stretching Exercise
Number analyzed (Participants) | 52 | 51
Days | 13 [10 to 18.5] | 17 [13 to 23]

ADVERSE EVENTS:
Time Frame: From enrollment to end of follow-up, up to 30 days.
Arm/Group | Aerobic Exercise | Stretching Exercise
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 0/52 | 0/51

LIMITATIONS AND CAVEATS:
Participants were not blinded to treatment; thus, intervention bias is possible. We think this unlikely, since all participants received an active intervention without being told which might be better, and they received equal attention from the investigators.We did not assess expectation of benefit (ie, perceived credibility of each intervention prior to initiation) to estimate the potential magnitude of expectancy bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT02710123/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT02710123/ICF_001.pdf